CLINICAL TRIAL: NCT01930565
Title: Comparison of Clinical and Histological Effects Between Lactobacillus Fermented Chamaecypris Obtusa and Tea Tree Oil for the Treatment of Mild to Moderate Acne: an 8-week Double Blind, Randomized Controlled, Split-face Study
Brief Title: Effectiveness and Safety of New Botanical Component-LFCO- Compared With Existing TTO in Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dae Hun Suh, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: H-1209-069-427
Record Dates: First submitted 2013-08-20; First posted 2013-08-29 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Acne Vulgaris
Keywords: acne; therapeutics; clinical trial; natural compound; Lactobacillus fermented Chamaecypris obtuse; tea tree oil
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LFCO application (Experimental): We made LFCO application(Lactobacillus Fermented Chamaecypris obtusa) containing cream to one side of patients' face to monitor effectiveness and safety in acne treatment.
  Interventions: Other: LFCO application
- TTO application (Active Comparator): To compare effectiveness and safety of new LFCO, we applied existing TTO containing cream to the other side of face in the same patients
  Interventions: Other: TTO application

INTERVENTIONS:
Other: LFCO application — Application of LFCO (Lactobacillus fermented Chamaecypris obtusa ) containing creams to one randomly selected face of patients to monitor its effectiveness and safety of acne treatments.
  Other Names: LFCO containg creams applied to acne lesions
  Arms: LFCO application
Other: TTO application — Application of TTO (Tea tree oil) containing creams to the other side of face of patients to monitor its effectiveness and safe compared with LFCO.
  Other Names: TTO containg creams applied to acne lesions
  Arms: TTO application

SUMMARY:
In an 8 week double blind randomized controlled split-face studies, we tried to compare the clinical efficacy, safety and histopathological changes between Lactobacillus fermented Chamaecypris obtusa (LFCO) and existing tea tree oil (TTO)

Basically, this is a split face study - one side of face randomly assigned was applied with LFCO and the other side with TTO in same patients.

DETAILED DESCRIPTION:
Screening of natural compounds for the development of anti-acne therapeutic agents has been steadily required considering various side effects of acne medications.However, previous studies have mainly focused on experimental tests without clinical trials and histopathological analysis.

To compare the clinical efficacy, safety and histopathological changes between Lactobacillus fermented Chamaecypris obtusa (LFCO) and existing tea tree oil (TTO)

Total thirty four patients were instructed to apply 5 % LFCO to the involved areas of randomly allocated side and 5 % TTO extract to the other side for 8 weeks in a double blind split-face clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* age 19-45
* active acne lesions in both sides of face
* available during study periods

Exclusion Criteria:

* pregnancy, mental illness, intake of oral isotretinoin within 6 months, application of the other oral or topical acne medications, chemical peeling or light based treatments within 6 weeks.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Number of inflammatory and non-inflammatory acne lesions | total 8 weeks after baseline
  Compared to baseline, number inflammatory and non-inflammatory acne lesions were counted to check out the effectiveness & safety of two botanical compounds

SECONDARY OUTCOMES:
Patient's subjective assessments for comfortableness & efficacy | 8 weeks after baseline
  Patients are required to report subjective assessments for comfortableness & efficacy for two creams they used
Sebum secretion assessment | 8 weeks after baseline
  Patients' sebum secretion from face was measured by sebumeter to detect sebum secretion changes after applying two components.
Histopathologic analysis | 8 weeks after baseline
  changes of tissue after application of two creams
Adverse effects | 8 weeks after baseline
  patients' reportings for severe side effects after application of two creams was monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hun Sun, MD, Study Chair — Seoul National University Hospital
Locations (1):
- Department of Dermatology, Seoul National University College of Medicine, Seoul, South Korea

REFERENCES:
- [Result] Hayashi N, Kawashima M. Multicenter randomized controlled trial on combination therapy with 0.1% adapalene gel and oral antibiotics for acne vulgaris: comparison of the efficacy of adapalene gel alone and in combination with oral faropenem. J Dermatol. 2012 Jun;39(6):511-5. doi: 10.1111/j.1346-8138.2011.01450.x. Epub 2011 Dec 14. PMID 22168326
- [Result] Enshaieh S, Jooya A, Siadat AH, Iraji F. The efficacy of 5% topical tea tree oil gel in mild to moderate acne vulgaris: a randomized, double-blind placebo-controlled study. Indian J Dermatol Venereol Leprol. 2007 Jan-Feb;73(1):22-5. doi: 10.4103/0378-6323.30646. PMID 17314442
- See also: Related Info — http://www.accessdata.fda.gov/scripts/cder/drugsatfda